CLINICAL TRIAL: NCT04624113
Title: Tazemetostat and Pembrolizumab in Patients With Pembrolizumab- or Nivolumab-Resistant, Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma: A Phase 1-2 Trial
Brief Title: Tazemetostat and Pembrolizumab in Patients With Pembrolizumab- or Nivolumab-Resistant, Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Ipsen bought out Epizyme
Sponsor: Washington University School of Medicine (Other)
Collaborators: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202011174
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tazemetostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: Tazemetostat + Pembrolizumab (Experimental): * Cycle 1 over 5 weeks (35 days). Subsequent cycles over 3 weeks (21 days).
  * Tazemetostat tablet twice per day Days 1-35 of Cycle 1, then Days 1-21 of subsequent cycles. Dose of tazemetostat will depend on dose level assigned
  * Pembrolizumab 200mg intravenous Day 15 of Cycle 1, then Day 1 of subsequent cycles.
  Interventions: Drug: Tazemetostat; Drug: Pembrolizumab
- Phase 2: Tazemetostat + Pembrolizumab (Experimental): * Cycle 1 over 5 weeks (35 days). Subsequent cycles over 3 weeks (21 days).
  * Tazemetostat tablet twice per day Days 1-35 of Cycle 1, then Days 1-21 of subsequent cycles. Dose of tazemetostat will depend of recommended phase 2 determined in Phase I portion of study.
  * Pembrolizumab 200mg intravenous Day 15 of Cycle 1, then Day 1 of subsequent cycles.
  Interventions: Drug: Tazemetostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Tazemetostat — Epizyme will supply the study agent, which will be provided free of charge to the patient.
  Other Names: Tazverik
Drug: Pembrolizumab — Pembrolizumab is commercially available
  Other Names: Keytruda

SUMMARY:
The primary aim of the phase 1 portion of the trial is to establish the recommended phase 2 dose (RP2D) of tazemetostat in combination with a fixed dose of pembrolizumab in patients with recurrent or metastatic (RM) head and neck cancer.

The primary aim of the phase 2 portion of the trial is to establish the proportion of patients with pembrolizumab- or nivolumab-resistant, PD-L1 positive, RM head and neck squamous-cell carcinoma (HNSCC) who achieve an objective tumor response to tazemetostat and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Phase 1 specific: recurrent or metastatic head and neck cancer, inclusive of cancers that originate in the head and neck, except central nervous system (CNS) cancers.
  * Phase 2 specific: recurrent or metastatic head and neck squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx.
* Disease Evaluation:

  * Phase 1 specific: Measurable or evaluable disease
  * Phase 2 specific: Measurable disease per RECIST. Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Phase 2 specific: Progression of disease, as assessed by RECIST, that occurred on prior pembrolizumab or nivolumab (given alone or with other therapy) in the last 6 months.
* Phase 2 specific: PD-L1 positive (CPS ≥ 1 by IHC, 22C3 antibody) on archived tumor tissue. If CPS not available, tumors with PD-L1 TPS ≥ 1 are also eligible (but CPS should be performed in these cases).
* Incurable disease (defined as surgery and/or radiation is unable to offer curative potential), or ineligible for (or patient declined) local therapy.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 750/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 9 g/L
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Serum creatinine <1.5x ULN or Creatinine clearance ≥ 50 mL/min by Cockcroft-Gault
* The effects of tazemetostat on the developing human fetus are unknown. For this reason and because histone methyltransferase (HMT) agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 6 months after the last day of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and for 6 months after last day of treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Radiation, chemotherapy, or targeted therapy within 14 days of treatment start.
* Phase 2 specific: Prior therapy with an EZH2 inhibitor.
* Investigational therapy within 21 days of treatment start.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 1 year before registration and the patient has no evidence of disease.
* Has known active CNS metastases. Subjects with previously treated brain metastases may participate provided they are stable (without any evidence of progression by imaging 4 weeks prior to the first dose of study treatment and any neurologic symptoms have stabilized), have no evidence of new or enlarging brain metastases, and are on stable or tapering doses of steroids for at least 14 days prior to first dose of study treatment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to tazemetostat, pembrolizumab, or other agents used in the study.
* Unable to swallow oral medication.
* Receiving systemic corticosteroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of treatment. A history of severe autoimmune disorder requiring high-dose corticosteroid treatment due to prior PD-1 inhibitor is an exclusion criterion.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of treatment.
* Prior organ or allogeneic stem cell transplant.
* Has an active autoimmune disease (i.e. rheumatoid arthritis, lupus, Sjogren's syndrome) that has required IV or subcutaneous systemic treatment in the past 6 months (excluding Rituxan). Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of tazemetostat in combination with a fixed dose of pembrolizumab (Phase I only) | Completion of cycle 1 for all phase I participants (estimated to be 9 months)
Objective response rate (ORR) assessed by iRECIST (Phase 2 only) | Through completion of treatment (estimated to be 5 months)
  -ORR: complete or partial response achieved as best response divided by those participants who have received a response evaluation (scan)

SECONDARY OUTCOMES:
Incidence of adverse events | From start of treatment through 28 days post-treatment (estimated to be 6 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Duration of response (DOR) | Through completion of treatment (estimated to be 5 months)
  -Response duration will be measured from the time measurement criteria for CR/PR or iCR/iPR (whichever is first recorded) are first met until the first date that recurrent or PD is objectively documented, taking as reference the smallest measurements recorded on study (including baseline).
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 17 months)
  -PFS is defined as the time from date of study enrollment to disease progression or death from any cause, whichever occurs first. The patients alive, without progression, are censored at the last follow-up.
Overall survival (OS) | Through completion of follow-up (estimated to be 17 months)
  -OS is defined as the time from the date of treatment to the date of death, censored at the last follow-up otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu